CLINICAL TRIAL: NCT01865682
Title: Effects of Varying Trim Lines of Solid Ankle-foot Orthoses on Ankle and Knee Kinematics and Kinetics During Stance Phase.
Brief Title: Effect of Ankle-foot Orthoses Trim Line Modifications on Ankle and Knee Motion and Force.
Status: Completed | Type: Observational
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Dana Craig, Health System Specialist, Southern California Institute for Research and Education
Other Study IDs: VALB-1215
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Lower Extremity Biomechanics
Keywords: Ankle; Knee; Orthosis; Kinematics; Kinetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to quantify changes in ankle and knee motion and force resulting from five progressive modifications to the anterior-posterior trim lines of thermoformed ankle-foot orthoses (AFO). It is hypothesized that the AFO with the most anterior trim line will prevent the most plantar flexion during loading response (the first 10% of the gait cycle)and prevent the most dorsiflexion at terminal stance (from 30 to 50% of the gait cycle) as compared to the non-device condition. This will be evidenced by the sagittal plane ankle motion and ground reaction force magnitude and location during loading response and terminal stance. Additionally, the angular velocity of knee flexion will increase during these same periods. By contrast, as the trim lines are moved more posterior this will result in lowering the effective stiffness of the device which will result in progressive increases in dorsiflexion and allow increasing amounts of knee flexion during terminal stance.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have no known pathology that would affect their ambulatory ability.
* Age greater than or equal to 18 years, but less than 40 years.
* Ability to tolerate walking for a minimum of 100 yards over the course of a three and a half hour time period.
* No current skin breakdown or sores on either lower extremity.

Exclusion Criteria:

* Use of ambulatory aids such as canes or crutches.
* Any medical or psychological condition that could jeopardize the subject's participation and compliance with the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study seeks to recruit younger, healthy (non-pathological) individuals over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sagittal plane ankle angle. | Six months

SECONDARY OUTCOMES:
Sagittal plane knee angle. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Dana D. Craig, MA, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Hsu, J., Michael, J., Fisk, J. (2008) AAOS Atlas of Orthoses and Assistive Devices. Mosby Inc., Elsevier, Inc. Pennsylvania
- [Background] Lusardi, M. and Nielsen, C.(2007) Orthotics and Prosthetics in Rehabilitation. Elsevier, Inc. Missouri
- [Background] White H, Jenkins J, Neace WP, Tylkowski C, Walker J. Clinically prescribed orthoses demonstrate an increase in velocity of gait in children with cerebral palsy: a retrospective study. Dev Med Child Neurol. 2002 Apr;44(4):227-32. doi: 10.1017/s0012162201001992. PMID 11995890
- [Background] Jagadamma KC, Owen E, Coutts FJ, Herman J, Yirrell J, Mercer TH, Van Der Linden ML. The effects of tuning an ankle-foot orthosis footwear combination on kinematics and kinetics of the knee joint of an adult with hemiplegia. Prosthet Orthot Int. 2010 Sep;34(3):270-6. doi: 10.3109/03093646.2010.503225. PMID 20738231
- [Background] Radtka SA, Skinner SR, Johanson ME. A comparison of gait with solid and hinged ankle-foot orthoses in children with spastic diplegic cerebral palsy. Gait Posture. 2005 Apr;21(3):303-10. doi: 10.1016/j.gaitpost.2004.03.004. PMID 15760746
- [Background] Desloovere K, Molenaers G, Van Gestel L, Huenaerts C, Van Campenhout A, Callewaert B, Van de Walle P, Seyler J. How can push-off be preserved during use of an ankle foot orthosis in children with hemiplegia? A prospective controlled study. Gait Posture. 2006 Oct;24(2):142-51. doi: 10.1016/j.gaitpost.2006.08.003. Epub 2006 Aug 24. PMID 16934470